CLINICAL TRIAL: NCT02785783
Title: Endorings™ Assisted Colonoscopy Versus Standard Colonoscopy for Polyp Detection in Symptomatic and Asymptomatic Patients: A Randomised Controlled Trial
Brief Title: Endorings™ Assisted Colonoscopy Versus Standard Colonoscopy for Polyp Detection
Acronym: Erings™
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Portsmouth Hospitals NHS Trust (Other Government)
Collaborators: University of Portsmouth (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: PHT/2015/101
Record Dates: First submitted 2016-05-25; First posted 2016-05-30 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Colorectal Neoplasia; Intestinal Neoplasms; Digestive Neoplasms; Digestive System Disease; Intestinal Disease; Gastrointestinal Disease; Gastrointestinal Neoplasm
Keywords: EndoRings™
MeSH Terms: conditions — Intestinal Neoplasms; Digestive System Diseases; Intestinal Diseases; Gastrointestinal Diseases; Gastrointestinal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard colonoscopy (Active Comparator): A standard colonoscope will be used to complete the procedure
  Interventions: Device: Standard colonoscopy
- EndoRings™ (Active Comparator): An EndoRings™ device will be placed at the distal end of a standard colonoscope
  Interventions: Device: EndoRings™

INTERVENTIONS:
Device: Standard colonoscopy
  Other Names: Current standard of care colonoscopy
  Arms: Standard colonoscopy
Device: EndoRings™ — Colonoscopy performed with an EndoRings™ device at the tip of a standard colonoscope
  Arms: EndoRings™

SUMMARY:
This study evaluates the impact of Endorings™ assisted colonoscopy on the number of polyps detected per patient compared to standard colonoscopy without use of EndoRings™. Half of the participants will receive EndoRings™ assisted colonoscopy, while the other half will receive standard colonoscopy.

DETAILED DESCRIPTION:
Colonoscopy is the gold standard for detection of colorectal neoplasia (polyps and cancers) but it is well known that colonoscopy is associated with a neoplasia miss rate of up to 25%.

One such method of reducing the neoplasia miss rate is cap assisted colonoscopy, where a cap is placed at the distal end of the colonoscope.The theory behind how the cap aids mucosal visualisation is that it depresses and flattens colonic folds, thereby improving visualisation on the proximal sides of folds.

Investigators aim to evaluate the impact of one such cap assisted device: EndoRings™ on polyp detection rates. EndoRings™ has been shown to improve polyp detection rate by 51% compared to 29% for standard colonoscopy in a recent tandem endoscopy study. EndoRings™ has received FDA approval.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic patients referred for colonoscopy age ≥ 55.
* Asymptomatic patients age ≥55 undergoing screening or surveillance for polyps and cancers.

Exclusion Criteria:

* History of Inflammatory bowel disease
* History of Hereditary non polyposis colorectal cancer (HNPCC)
* Familial adenomatous polyposis syndrome (FAP)
* Hyperplastic polyposis syndrome
* Known colonic stricture

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 563 (Actual)
Dates: Start 2016-05-13 (Actual); Primary Completion 2018-08-07 (Actual); Study Completion 2018-08-07 (Actual)

PRIMARY OUTCOMES:
Number of polyps per patient | 14 months
  To assess the impact of the Endorings™ cap on the number of polyps detected per patient as compared to standard colonoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Pradeep Bhandari, MD, Principal Investigator — Portsmouth University Hospital
Locations (1):
- Portsmouth University Hospital, Portsmouth, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Rijn JC, Reitsma JB, Stoker J, Bossuyt PM, van Deventer SJ, Dekker E. Polyp miss rate determined by tandem colonoscopy: a systematic review. Am J Gastroenterol. 2006 Feb;101(2):343-50. doi: 10.1111/j.1572-0241.2006.00390.x. PMID 16454841
- [Background] Dik VK, Gralnek IM, Segol O, Suissa A, Belderbos TD, Moons LM, Segev M, Domanov S, Rex DK, Siersema PD. Multicenter, randomized, tandem evaluation of EndoRings colonoscopy--results of the CLEVER study. Endoscopy. 2015 Dec;47(12):1151-8. doi: 10.1055/s-0034-1392421. Epub 2015 Jul 28. PMID 26220283